CLINICAL TRIAL: NCT00977613
Title: Prospective Evaluation of Adherence to Recommended Activity Regimen in Patients Following Treatment of Stages II and III Colorectal Cancer.
Brief Title: Adherence to a Recommended Exercise Regimen in Colorectal Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Medical Center (Other)
Responsible Party: Peter Kozuch, MD, Beth Israel Medical Center
Allocation: Not Applicable | Model: Single Group
Other Study IDs: 003-07
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Results first posted 2011-02-28 (Estimated); Last update posted 2011-03-03 (Estimated); Status verified 2011-03

CONDITIONS: Colorectal Cancer (CRC)
Keywords: Treated Stage 2 and Stage 3 colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- life style counseling (Other): Treated stage 2 and 3 colorectal cancer patients were counseled to exercise at least to the equivalent of 18 metabolic hours per week and were assessed over 6 months.
  Interventions: Behavioral: exercise counseling

INTERVENTIONS:
Behavioral: exercise counseling — motivational counseling to exercise a minimum 18 metabolic hours per week

SUMMARY:
Given the apparent effect of 18 metabolic equivalent task-hours of activity/week in improving disease free survival in patients with treated stage 3 colon cancer and the survival benefit of exercise demonstrated in patients with stage II and III colorectal cancer, the primary objective is to evaluate compliance at 6 months with post-treatment recommendations for a minimum of 18 metabolic units of physical activity each week in patients who have completed therapy for stage 2 and stage 3 colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histological confirmation of stage 2 or stage 3 colorectal cancer.
2. Ability to sign written informed consent.
3. WHO performance status of 2 or better.
4. No evidence of recurrent disease or death prior to second questionnaire.
5. Patients with declining physical activity within 90 days of second physical activity assessment will be excluded.

There are no exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-04; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Kozuch, MD, Principal Investigator — Beth Israel Medical Center
Locations (2):
- United States (2):
  - Beth Israel Medical Center - Philipps Ambulatory Care Center, New York, New York
  - St. Luke's Roosevelt Hospital Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolled subjects were ambulatory patients completing treatment for colorectal cancer (CRC) from April 2007 through August 2009 at the Continuum Cancer Centers-Beth Israel Medical Center and St. Luke's Roosevelt Hospital.
Pre-assignment Details: Subjects were counseled to exercise at least 18 metabolic equivalent units weekly. Subjects were provided with information on the metabolic equivalents of common forms of exercise.
Groups:
- Single Arm, Life Style Counseling: Patients with stage II or III colon or rectal cancer were accrued by physician screening at a visit three to four months following surgical resection. At the time of initial subject study enrollment, and at each follow-up visit, the physician or nurse administering the questionnaire was to review the benefit of adjuvant exercise and encourage patients to continue or increase their weekly activity in order to maintain at least 18 MET/week.
Period: Overall Study
Arm/Group | Single Arm, Life Style Counseling
Started | 50
Completed | 34
Not Completed | 16
Not completed — Lost to Follow-up | 16

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm, Life Style Counseling
Number analyzed (Participants) | 50
Age, Customized [Number; unit: participants]
  Age greater than 18 years | 50
Sex/Gender, Customized [Number; unit: participants]
  Female | 21
  Male | 26
  Unknown | 3
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Maintained an Exercise Regimen Average of 18 Metabolic Units (MET) Per Week or Greater
Description: One MET is the energy expenditure for sitting quietly for 1 hour. MET scores for walking were assigned based on the pace and duration reported. For other activities, a leisurely to moderate intensity score was selected. The scores for MET-hours per week for each activity were calculated from the reported hours per week engaged in that activity multiplied by the assigned MET score, and individual activities were summed to derive a total MET-hours per week.
Time Frame: 6 months
Population: 34 of the 50 enrolled subjects had at least 6 months of follow-up. There was no evaluable data for the remaining 16 subjects.
Measure: Number; unit: participants
Arm/Group | Single Arm, Life Style Counseling
Number analyzed (Participants) | 34
participants | 18

2. Secondary Outcome: Disease-free Survival
Time Frame: after 6 months
Reporting Status: Not Posted

3. Secondary Outcome: Recurrence-free Survival
Time Frame: after 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Overall Survival
Time Frame: after 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Single Arm, Life Style Counseling
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

LIMITATIONS AND CAVEATS:
Many participants were lost to follow-up. Some participants had not been followed for at least 6 months at study termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes